CLINICAL TRIAL: NCT00171886
Title: Octreotide Efficacy and Safety in First-line Acromegalic Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSMS995BES02
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2011-03

CONDITIONS: Acromegaly
Keywords: Acromegaly; Otreotide; Tumor reduction
MeSH Terms: conditions — Acromegaly | interventions — Octreotide

ARMS (1):
- octrotide (Experimental)
  Interventions: Drug: Octreotide

INTERVENTIONS:
Drug: Octreotide
  Other Names: SMS995

SUMMARY:
Primary Acromegaly is a clinical and metabolic disease caused by growth hormone (GH) hypersecretion from a pituitary adenoma and is an insidious, chronic disease that is associated with bony and soft tissue overgrowth. Goals of therapy are to eradicate the tumor, suppress GH secretion, normalize IGF-I levels, and preserve normal pituitary function.

This study will evaluate the safety and efficacy of octreotide as primary therapy for the treatment of acromegaly and as therapy for patients with acromegaly and a pituitary macroadenoma or microadenoma.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 18 and < 80 years old.
* Recently diagnosed not previously treated patients with acromegaly.
* Presence of a pituitary tumor (microadenoma or macroadenoma), documented by a MNR performed in the 12 weeks before enrolment.
* Absence of nadir suppression of the nadir of GH to < 1.0 ng/mL, after oral administration of 75 g of glucose (OTTG).
* IGF-I levels over normal upper limits, e.g. 97 percentile (age- and sex-matched).
* Tolerance shown with a test of a subcutaneous injection of octreotide
* Written Informed Consent before any procedure specific to the study. Inclus

Exclusion Criteria:

* Previously treated patients with any therapy for acromegaly, including surgery, radiotherapy, bromocriptin, and somatostatin analogues.
* Compression of optic chiasm that produces any impairment of field of vision.
* Need of surgery to improve any neurological sign or symptom associated with a direct incidence on the tumour.
* Intolerance to octreotide or to any component of Sandostatin® LAR® preparation.
* Patients with an hepatic condition such as cirrhosis, active or persisting chronic hepatitis, or other hepatopathy of fast evolution.
* Pregnant women
* History of alcohol or drug abuse in the six months prior to the inclusion visit.
* Patients suffering from any condition that may jeopardize the interpretation of study results or may impede to obtain informed consent
* Intake of an investigational drug during the study and 30 days before patient inclusion in this study

Other protocol-defined inclusion / exclusion criteria may apply.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2002-07; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
To evaluate the ability of Sandostatin® LAR® to decrease GH and IGF-I levels in acromegaly patients with micro- or macroadenomas not previously treated | at baseline, weeks 12, 24, 48
To evaluate efficacy of Sandostatin® LAR® to reduce the size of micro- or macroadenomas in acromegaly patients with micro- or macroadenomas not previous treated | at baseline, weeks 12, 24, 48

SECONDARY OUTCOMES:
To evaluate the effect of Sandostatin® LAR® on Health Related Quality of Life. | at baseline, weeks 12, 24, 48
To evaluate the ability of Sandostatin® LAR® to relieve acromegaly signs and symptoms | at baseline, weeks 12, 24, 48

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (8):
- Spain (8):
  - Novartis Investigative site, A Coruña
  - Novartis Investigative site, Alicante
  - Novartis Investigative site, Barcelona
  - Novartis Investigative site, Burgos
  - Novartis Investigative site, Córdoba
  - Novartis Investigative site, Madrid
  - Novartis Investigative site, Málaga
  - Novartis Investigative site, Tarragona